CLINICAL TRIAL: NCT04961268
Title: Effect of Preoperative Oral Tramadol on the Anaesthetic Efficacy of Inferior Alveolar Nerve Block in Patients With Symptomatic Irreversible Pulpitis: A Prospective, Randomized, Double-blind, Controlled Study
Brief Title: Effect of Preoperative Oral Tramadol on Inferior Alveolar Nerve Block in Patients With Symptomatic Irreversible Pulpitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alfarabi Colleges (Other)
Responsible Party: Principal Investigator, Amr Elnaghy, Associate Professor, Alfarabi Colleges
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Alfarabi
Record Dates: First submitted 2021-07-01; First posted 2021-07-14 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Symptomatic Irreversible Pulpitis
Keywords: anaesthesia; endodontics; inferior alveolar nerve block; NSAIDs; tramadol
MeSH Terms: interventions — Tramadol; Tablets; Ibuprofen; Acetaminophen

STUDY DESIGN:
Intervention Model Description: The study included five study groups, each consists of 50 patients who exhibited symptomatic irreversible pulpitis of a mandibular first or second molar. The patients received identically appearing capsules containing either tramadol 50 mg, tramadol 100 mg, ibuprofen 600 mg, ibuprofen 600 mg/acetaminophen 1000 mg or placebo by mouth 60 min before the administration of an IANB. Endodontic access was begun 15 min after completion of the IANB, and all patients used for data analysis had profound lip numbness. The IANB success was defined as no or mild pain (visual analog scale recordings) on pulpal access or instrumentation.
Who Masked: Participant, Investigator
Masking Description: To blind the experiment, each of the 50 patients in each group was randomly allocated a code consists of 2 letters and one number. Only the random numbers identified the medications; thus, the patient and doctor were uninformed of which medication was given to them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Tramadol 50 (Active Comparator): Before the inferior alveolar nerve block injection by 60 minutes, the patient received tramadol 50 mg in opaque yellow size "000" capsules.
  Interventions: Drug: TraMADol 50 Mg Oral Tablet
- Tramadol 100 (Active Comparator): Before the inferior alveolar nerve block injection by 60 minutes, the patient received tramadol 100 mg in opaque yellow size "000" capsules.
  Interventions: Drug: Tramadol 100 MG Oral Tablet
- Ibuprofen (Active Comparator): Before the inferior alveolar nerve block injection by 60 minutes, the patient received ibuprofen 600 mg in opaque yellow size "000" capsules.
  Interventions: Drug: Ibuprofen 600Mg Tab
- Ibuprofen/acetaminophen (Active Comparator): Before the inferior alveolar nerve block injection by 60 minutes, the patient received ibuprofen 600 mg/acetaminophen 1000 mg in opaque yellow size "000" capsules.
  Interventions: Drug: ibuprofen 600 mg/acetaminophen 1000 mg
- Placebo (Placebo Comparator): Before the inferior alveolar nerve block injection by 60 minutes, the patient received Placebo in opaque yellow size "000" capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TraMADol 50 Mg Oral Tablet — The patients were randomly given the medication by mouth 60 min before administering IANB.
  Other Names: TRAMAL
  Arms: Tramadol 50
Drug: Tramadol 100 MG Oral Tablet — The patients were randomly given the medication by mouth 60 min before administering IANB.
  Other Names: TRAMAL
  Arms: Tramadol 100
Drug: Ibuprofen 600Mg Tab — The patients were randomly given the medication by mouth 60 min before administering IANB.
  Other Names: IBUPROFEN
  Arms: Ibuprofen
Drug: ibuprofen 600 mg/acetaminophen 1000 mg — The patients were randomly given the medication by mouth 60 min before administering IANB.
  Other Names: IBUPROFEN/PANADOL
  Arms: Ibuprofen/acetaminophen
Drug: Placebo — The patients were randomly given the medication by mouth 60 min before administering IANB.
  Arms: Placebo

SUMMARY:
Aim: The purpose of this prospective, randomized, double-blind, controlled study was to compare the preoperative oral tramadol medication with ibuprofen and acetaminophen on the success of inferior alveolar nerve blocks (IANB) of mandibular posterior teeth in patients experiencing symptomatic irreversible pulpitis.

Methodology: The study included five study groups, each consists of 50 patients who exhibited symptomatic irreversible pulpitis of a mandibular first or second molar. The patients received identically appearing capsules containing either tramadol 50 mg, tramadol 100 mg, ibuprofen 600 mg, ibuprofen 600 mg/acetaminophen 1000 mg or placebo by mouth 60 min before the administration of an IANB. Endodontic access was begun 15 min after completion of the IANB, and all patients used for data analysis had profound lip numbness. The IANB success was defined as no or mild pain (visual analog scale recordings) on pulpal access or instrumentation. The data were analysed using chi-square χ2 and Kruskal-Wallis tests.

DETAILED DESCRIPTION:
This study was designed as a double-blind, randomized, placebo-controlled clinical trial. This trial was carried out according to the latest update of the Declaration of Helsinki guidelines (October 2013) and approved by the Vision Colleges Research Ethics Committee (approval number 20-5/2). The patients were pre-selected to participate based on a preoperative pain scale of preliminary clinical assessment following the guidelines suggested by the CONSORT group for planning and reporting clinical trials. A total of 275 adult patients were screened for participation in this study. They were emergency patients of the Vision Colleges Dental Clinics and were in good health based on their medical histories and oral questioning. Subjects who were less than 18 years old, had a history of serious medical problems, had used central nervous system depressants or any analgesic medication within the previous 6 hours, were pregnant or were unable to give informed consent were all excluded from the study. Finally, 50 patients were enrolled in each group, for a total of 250 patients.

The inclusion criteria were active pain in a mandibular molar first or/and the second molar, prolonged response to cold testing (Endo-frost; Roeko, Langenau, Germany), absence of any periapical radiolucency on periapical radiographs, and a vital coronal pulp on access opening. The Modified Dental Anxiety Scale assessed the level of anxiety among the patients. The pain of the patients was categorized into four categories using the Heft-Parker visual analogue scale (HP VAS):

0 mm: no pain 0-54 mm: faint, weak, or mild 55-114 mm: moderate pain >114 mm: strong, intense, and maximum possible All patients were randomly divided using block randomisation to ensure the homogeneity of the five groups. The patients were randomly given tramadol 50 mg, tramadol 100 mg, ibuprofen 600 mg, ibuprofen 600 mg/acetaminophen 1000 mg or placebo by mouth 60 min before administering IANB. To blind the experiment, each of the 50 patients in each group was randomly allocated a code consists of 2 letters and one number. Only the random numbers identified the medications; thus, the patient and doctor were uninformed of which medication was given to them. The medication and placebo were blinded in the following way. In opaque yellow size "000" capsules, a certified pharmacist prepared identical-appearing capsules of the medications and placebo in identical separate containers for each medication. At 60 minutes after receiving the medication or placebo, the operator used a cotton tip applicator to put anaesthetic gel (20 percent benzocaine; Patterson Dental Supply, Inc, St Paul, MN, USA) at the IANB injection site for 60 s.

The participants were then given regular IANB injections and 0.9 mL long buccal injections containing 2% lidocaine and 1:100,000 epinephrine (Xylocaine; Astra Zeneca LP, Dentsply, York, PA, USA). The first author used self-aspirating syringes (Septodont, Sant-Maur-des-Fosses Cedex, France) and 27-G long needles to inject the anaesthetic solution (Septoject, Septodont). Each patient was asked for lip numbness every 5 min for 15 min after the IANB. The block was considered missed if substantial lip numbness was not reported by 15 min, and the participant was excluded from the trial. Due to a lack of lip numbness, no patients were excluded.

After that, a rubber dam was used to isolate the teeth and endodontic access was conducted. During the endodontic process, patients were asked to rate any pain they experienced. If the patient was in pain, the treatment was stopped, and the patient used the HP VAS to rate his/her discomfort. The success of the IANB was defined as the ability to access and clean and shape the tooth without pain (VAS score of 0) or mild pain (VAS rating ≤54 mm). The rubber dam was removed if the patient had moderate or severe pain (VAS rating ≥ 55 mm), and a buccal infiltration of a cartridge containing 4% articaine with 1:100,000 epinephrine (Septocaine; Septodont) was administrated buccally to the tooth that required emergency treatment. After 5 min, the rubber dam was replaced, and endodontic access was continued. The success of the buccal infiltration was defined as the ability to access and instrument the tooth without pain (VAS score of 0) or with mild pain (VAS rating ≤54 mm). Intraosseous anaesthesia was administrated to the patients who still had moderate to severe pain. The intraosseous injection was administrated with the Stabident intraosseous anaesthetic system (Fairfax Dental Inc, Miami, Fl, USA) using a cartridge of 2% lidocaine with 1:100,000 epinephrine as described previously. If that was not successful, an intrapulpal injection was given, and endodontic debridement was completed. The extent of access preparation and/or instrumentation was recorded as within dentine, within pulp space, and instrumentation of canals.

The VAS satisfaction form was used to record the post-treatment satisfaction of the patient. The patient was asked to draw a vertical line on the VAS (0-100 mm) to indicate their satisfaction with the entire treatment. The VAS was classified into four categories; 0: not satisfied, >0 mm and ≤33 mm: somewhat satisfied, >33 mm but <66 mm: moderately satisfied and ≥66 mm: completely satisfied.

Data of the study were collected and statistically analysed (SPSS 22.0 software; IBM Corp., Armonk, NY, USA) using chi-square χ2 test to compare between different groups for anaesthetic success, gender, and tooth type. Normality of data was tested by Shapiro-Wilk test. The Modified Dental Anxiety Scale, age, and initial pain ratings were analysed by using Kruskal-Wallis test. The level of statistical significance was set at P < 0.05. GPower v3.1.3 software (University of Düsseldorf; Düsseldorf, Germany) was used to calculate the sample size. According to a power analysis, a sample size of 50 patients per group meets the constraints of 0.05 and power = 0.95.

ELIGIBILITY:
Inclusion Criteria:

* active pain in a mandibular molar first or/and the second molar
* prolonged response to cold testing
* absence of any periapical radiolucency on periapical radiographs
* vital coronal pulp on access opening
* able to give informed consent

Exclusion Criteria:

* less than 18 years old
* history of serious medical problems
* used central nervous system depressants or any analgesic medication within the previous 6 hours
* pregnancy
* inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Pain Measurement as Assessed on a Heft-Parker 170 mm Visual Analog Scale | 15 minutes after the inferior alveolar nerve block.
  At 60 minutes after receiving the medication or placebo, the participants were then given inferior alveolar nerve block injection. Each patient was asked for lip numbness every 5 minutes for 15 minutes after inferior alveolar nerve block injection. During the endodontic process, patients were asked to rate any pain they experienced on a Heft-Parker visual analog scale. The number of millimeters along the scale were reported. No pain corresponded to 0 mm. Mild pain was defined as greater than 0 mm and less than or equal to 54 mm. Mild pain included the descriptors of "faint", "weak", and "mild pain". Moderate pain was defined as greater than 54 mm and less than 114 mm and included the descriptor "moderate". Severe pain was defined as equal to or greater than 114 mm up to and including 170 mm. Severe pain included the descriptors of "strong", "intense", and "maximum possible."

SECONDARY OUTCOMES:
Postoperative Satisfaction on a 100 mm Visual Analog Scale | Immediately post-procedure on Day 0
  Patients were rate their level of satisfaction after treatment procedure using a visual analog scale. The scale ranges from "not satisfied," to "somewhat satisfied," to "moderately satisfied," to "completely satisfied." Not satisfied corresponded to 0 mm. Somewhat satisfied was defined as greater than 0 mm and less than or equal to 33 mm. Moderately satisfied was defined as greater than 33 mm and less than 66 mm. Completely satisfied was defined as equal to or greater than 66 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Amr M Elnaghy, PhD, Principal Investigator — Associate Professor of Endodontics
Locations (1):
- Vission Colleges, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this study, after deidentification (text, tables, and figures).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: For individual participant data meta-analysis

REFERENCES:
- [Background] Argueta-Figueroa L, Arzate-Sosa G, Mendieta-Zeron H. Anesthetic efficacy of articaine for inferior alveolar nerve blocks in patients with symptomatic versus asymptomatic irreversible pulpitis. Gen Dent. 2012 Jan-Feb;60(1):e39-43. PMID 22313992
- [Background] Pulikkotil SJ, Nagendrababu V, Veettil SK, Jinatongthai P, Setzer FC. Effect of oral premedication on the anaesthetic efficacy of inferior alveolar nerve block in patients with irreversible pulpitis - A systematic review and network meta-analysis of randomized controlled trials. Int Endod J. 2018 Sep;51(9):989-1004. doi: 10.1111/iej.12912. Epub 2018 Mar 24. PMID 29480930
- [Background] Aggarwal V, Singla M, Kabi D. Comparative evaluation of effect of preoperative oral medication of ibuprofen and ketorolac on anesthetic efficacy of inferior alveolar nerve block with lidocaine in patients with irreversible pulpitis: a prospective, double-blind, randomized clinical trial. J Endod. 2010 Mar;36(3):375-8. doi: 10.1016/j.joen.2009.11.010. PMID 20171350
- [Background] Aggarwal V, Singla M, Miglani S. Comparative Evaluation of Anesthetic Efficacy of 2% Lidocaine, 4% Articaine, and 0.5% Bupivacaine on Inferior Alveolar Nerve Block in Patients with Symptomatic Irreversible Pulpitis: A Prospective, Randomized, Double-blind Clinical Trial. J Oral Facial Pain Headache. 2017 Spring;31(2):124-128. doi: 10.11607/ofph.1642. PMID 28437508
- [Background] Fowler S, Drum M, Reader A, Beck M. Anesthetic Success of an Inferior Alveolar Nerve Block and Supplemental Articaine Buccal Infiltration for Molars and Premolars in Patients with Symptomatic Irreversible Pulpitis. J Endod. 2016 Mar;42(3):390-2. doi: 10.1016/j.joen.2015.12.025. Epub 2016 Jan 28. PMID 26831048
- [Background] Yadav M, Grewal MS, Grewal S, Deshwal P. Comparison of Preoperative Oral Ketorolac on Anesthetic Efficacy of Inferior Alveolar Nerve Block and Buccal and Lingual Infiltration with Articaine and Lidocaine in Patients with Irreversible Pulpitis: A Prospective, Randomized, Controlled, Double-blind Study. J Endod. 2015 Nov;41(11):1773-7. doi: 10.1016/j.joen.2015.06.008. Epub 2015 Sep 26. PMID 26410153
- [Background] Lapidus D, Goldberg J, Hobbs EH, Ram S, Clark GT, Enciso R. Effect of premedication to provide analgesia as a supplement to inferior alveolar nerve block in patients with irreversible pulpitis. J Am Dent Assoc. 2016 Jun;147(6):427-37. doi: 10.1016/j.adaj.2016.01.006. Epub 2016 Mar 4. PMID 26952243
- [Background] Rogers BS, Botero TM, McDonald NJ, Gardner RJ, Peters MC. Efficacy of articaine versus lidocaine as a supplemental buccal infiltration in mandibular molars with irreversible pulpitis: a prospective, randomized, double-blind study. J Endod. 2014 Jun;40(6):753-8. doi: 10.1016/j.joen.2013.12.022. Epub 2014 Feb 8. PMID 24862701
- [Background] Fullmer S, Drum M, Reader A, Nusstein J, Beck M. Effect of preoperative acetaminophen/hydrocodone on the efficacy of the inferior alveolar nerve block in patients with symptomatic irreversible pulpitis: a prospective, randomized, double-blind, placebo-controlled study. J Endod. 2014 Jan;40(1):1-5. doi: 10.1016/j.joen.2013.09.009. Epub 2013 Oct 27. PMID 24331983